CLINICAL TRIAL: NCT07267273
Title: Effect of Betamethasone Phonophoresis in Treatment of Vitiligo
Brief Title: Betamethasone Phonophoresis For Vitiligo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ola sabry Abd-Elmaksoud tarabya, Resident at Physical Therapy for Surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Treatment of Vitiligo
Record Dates: First submitted 2025-11-23; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Beclomethasone; Phonophoresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients Group (Active Comparator): This group of patients composed of 30 Male and female patients who received betamethasone cream then after 20 minutes ultrasound was applied, three times per week for 1 month.
  Interventions: Drug: Beclomethasone
- Control Group (Active Comparator): This group of patients composed of 30 Male and female patients who received ultrasound then after 20 minutes patients received betamethasone cream, three times per week for 1 month.
  Interventions: Drug: Beclomethasone

INTERVENTIONS:
Drug: Beclomethasone — to determine the effect of betamethasone phonophoresis on vitiligo patients.
  Other Names: phonophoresis

SUMMARY:
Vitiligo is a skin disorder that results in the formation of depigmented patches or hypopigmented macules due to selective destruction or reduction of melanocytes the cells that produce pigment in our skin.

Vitiligo affects 0.1-2% of the World's population. People of all skin types and all ages can be affecte. In most of the cases, white patches develop or expand slowly overtime, and in some cases it never progress and remains stable . Vitiligo can be segmental or non-segmental depending upon the morphology of the clinical involvement. It can also be classified as stable or unstable based on the activity of disease.

Steroids act as anti-inflammatory and immunosuppressant agents. Even if different classes of steroids are now available, the mid- potent ones (e.g. betamethasone dipropionate 0.05% cream, 0.05% clobetasol propionate ointment) are usually preferred for the treatment of young patients .

Now days, topical corticosteroids are the most commonly prescribed agents in treatment of dermatologic conditions .Almost all treatments of vitiligo have borrowed from therapies whose prime targets have been another disease.

DETAILED DESCRIPTION:
Many theories have been put forward to explain the pathogenesis of vitiligo and mechanisms that leads to the loss of functional melanocytes from the epidermis. The important ones include a genetic predisposition, autoimmune destruction of melanocytes, altered redox status and free radical mediated melanocyte damage, heightened sympathetic response and catecholamines/neurotransmitter mediated melanocyte damage, and impaired melanocyte adhesion or melanocytorrhagy.Mode of therapy is based on decreasing the activity, thereby achieving stability and later inducing pigmentation.

Vitiligo is classified into Segmental Vitiligo, Non-Segmental Vitiligo and Unclassified according to Vitiligo Global Issues Consensus Conference.Segmental vitiligo lesions are characterized by generally one and less commonly two or multiple segments. Most common form is Uni-segmental form which consists of one or more macules particularly on one side of the body with the involvement of body hair with early age of onset, and rapid stabilization while non-segmental vitiligo lesions are distributed bilaterally in an acrofacial pattern (i.e. affecting the face, hands or feet) or scattered symmetrically over the entire body .

Non-segmental vitiligo (NVS) comprises of acrofacial, generalized, universal, mixed forms. NVS can initially have an acrofacial distribution, which can later progress to the generalized or universal form. Acrofacial vitiligo can affect face, hands and feet and generally involve the perioral region and tips of the fingers. In a study of latent class analyses, two types of non-segmental vitiligo have been identified; the first is of early onset (i.e. before the 12 years of age) and generally associated with halo naevus with premature greying of hair, while second type is of late onset and is mostly associated with an acrofacial pattern. In generalized vitiligo, patient had a few acrofacial lesions for 10 years that evolved within 6 months into generalized form, spreading to the trunk. Universal Vitiligo affects about 80-90% of body surface area and is the most common form of vitiligo.

Generalized vitiligo usually precedes Universal vitiligo. Mixed vitiligo is defined as the combined involvement of both segmental and non-segmental vitiligo in one patient. Generally segmental vitiligo precedes the non-segmental vitiligo. Rare class is also considered as Un-classified type and consists of Follicular Vitiligo, Vitiligo Punctate and Vitiligo Minor. Vitiligo minor is likely to be limited to dark skinned individuals. The term minor here refers to incomplete pigmentation with pale skin compared with healthy skin .

The presence of focal lesions (i.e., small isolated white macule) with no segmental distribution that have not evolved into non-segmental or segmental vitiligo after 1-2 years but can evolve to segmental vitiligo or non-segmental vitiligo is regarded as unclassifiable vitiligo .

In many instances, the first line therapy for vitiligo is topical medicaments. Regarding topical therapy that might be effective in treatment of vitiligo, topical corticosteroids are the usual first line treatment .

The ease of application, high rate of compliance, and low cost are the advantages of topical corticosteroid therapy for vitiligo .Several stronger corticosteroids are now available since their first introduction. They are used as monotherapy or in combination with other agents for increasing efficacy.Topical corticosteroids have been indicated and used during the last three decades for treatment of limited area of vitiligo.

Phonophoresis (PH) is the process of increasing skin absorption and penetration of the topical medications to the deep tissues using US. Topically applied drugs therapeutic effects depend on different factors such as rate, amount, drug penetration dept of the skin and the potential drug toxicological hazards on the tissues

Phonophoresis, also known as sonophoresis, has been claimed to enhance the percutaneous absorption of certain pharmacological agents such as anti- inflammatory steroids and local anesthetics from intact skin into the underlying subcutaneous structures by ultrasound, therefore improving their effectiveness. This procedure is commonly used in physical therapy practices. The procedure generally utilizes an ultrasound apparatus that generates frequencies of 0.7 to 1.1 MHz . The ultrasound intensities employed usually range from 0.0 to 3.0 Watts per cm2. Both continuous-mode as well as pulse-mode applications were utilized, and most treatments lasted from 5 to 8 mins, with the exception of treatments of larger areas (greater than 36 cm2) requiring more than 8 mins.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients diagnosed with vitiligo.
* Medically and psychologically stable patients.
* Good cognitive abilities to understand the requirements of the study.
* All patients enrolled to the study will have their informed consent.
* they had no contraindications to the use of therapeutic ultrasound

Exclusion Criteria:

* Pregnancy or lactation.
* Immunosuppression.
* Alcohol abuse.
* History of spontaneous re-pigmentation of lesions.
* Presence of skin characteristics that may interfere with study assessment.
* Active bacterial/viral infection.
* Patients on other immune suppressants and phototherapy
* Patients currently participating in any other clinical study
* Uncooperative patients.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
vitiligo Management | 3 Months
  Evaluation of the patients whom suffering from vitiligo and using betamethasone phonophoresis for the treatment of vitiligo using Vitiligo noticeability scale (VNC)

CONTACTS AND LOCATIONS:
Overall Officials: Nisreen Afify Abd-Elrasheed, Professor, Study Chair — Physical Therapy for Surgery,Faculty of Physical Therapy,Cairo University
Locations (1):
- Cairo University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
No IPD sharing as participants request